CLINICAL TRIAL: NCT03035734
Title: A Randomized Study to Evaluate the Bioavailability of BMS-986141 From a Form B Tablet Formulation Relative to the Form A Reference Tablet in Healthy Participants
Brief Title: Evaluate the Bioavailability Between 2 BMS-986141 Formulations in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV006-023; 2016-001031-13 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2017-01-30 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Active Comparator): Single oral dose BMS-986141 Form A tablet under fasting conditions
  Interventions: Drug: BMS-986141 Form A Tablet
- B (Experimental): Single oral dose BMS-986141 Form B tablet (low-dose) under fasting conditions
  Interventions: Drug: BMS-986141 Form B tablet (low dose)
- C (Experimental): Single oral dose BMS-986141 Form B tablet (high-dose) under fasting conditions
  Interventions: Drug: BMS-986141 Form B tablet (high dose)
- D (Experimental): Single oral dose BMS-986141 Form B tablet (high-dose) under fed conditions
  Interventions: Drug: BMS-986141 Form B tablet (high dose)

INTERVENTIONS:
Drug: BMS-986141 Form A Tablet — tablet
  Arms: A
Drug: BMS-986141 Form B tablet (low dose) — tablet
  Arms: B
Drug: BMS-986141 Form B tablet (high dose) — tablet
  Arms: C; D

SUMMARY:
Open label, randomized, 4-period crossover study with single doses of BMS-986141 given to healthy female subjects of non-childbearing potential and healthy males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by no significant deviations in normal medical and surgical history and assessments
* Body mass index 18.0 kg/m2 to 32.0 kg/m2
* females must be of non-childbearing potential

Exclusion Criteria:

* known bleeding or coagulation disorders
* acute or chronic medical illness
* history of nausea or chronic diarrhea that lasts over 4 weeks
* history of periodontal disease or gingivitis which required treatment
* other exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the bioavailability between BMS-986141 Form B tablet compared to the Form A reference tablet | 4 weeks

SECONDARY OUTCOMES:
Further characterize safety and tolerability of BMS-986141 by assessing adverse events and other physical assessments throughout study conduct | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator inquiry form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx